CLINICAL TRIAL: NCT04606303
Title: A Single-center, Prospective, Single-arm Phase Ⅱ Trial of Neoadjuvant Toripalimab Plus Platinum-doublet Chemotherapy in Locally Advanced NSCLC.
Brief Title: A Phase Ⅱ Trial of Neoadjuvant Toripalimab Plus Platinum-doublet Chemotherapy in Locally Advanced NSCLC.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Wu Nan, Head of Department, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-DN-028
Record Dates: First submitted 2020-10-20; First posted 2020-10-28 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Locally Advanced NSCLC

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab Combined With Platinum-containing Dual-agent. (Experimental): Toripalimab combined with platinum-containing dual-agent as a neoadjuvant Therapy for Non-small Cell Lung Cancer.
  Interventions: Drug: Toripalimab combination with platinum-containing dual-drug chemotherapy.

INTERVENTIONS:
Drug: Toripalimab combination with platinum-containing dual-drug chemotherapy. — cisplatin + paclitaxel/ albumin-bound paclitaxel/ gemcitabine/ Pemetroxel+ Toripalimab (cisplatin 75mg/m2 (D1), paclitaxel 175mg/m2 (D1), or albumin-bound paclitaxel 260mg/m2 (D1), or gemcitabine 1250mg/m2 (D1, D8), or Pemetroxel 500mg/m2 (D1)), Toripalimab 240mg D1, Q3W.
  If the patient is SD or PD, Toripalimab combined with platinum-containing dual-drug chemotherapy in the third cycle will continue, and a total of 4 cycles can be carried out at most, and the therapeutic effect will be evaluated after each cycle of treatment. If the patient is PR or CR at any time during the treatment (after treatment in the third or fourth cycle), the surgical treatment will be entered. If PR or CR is still not reached after treatment in the fourth cycle, the endpoint of the trial will be reached, theobservation of the patient will be finished, and the subsequent treatment will be decided by the clinician.

SUMMARY:
This is a Phase 2, prospective, single-arm, open-Label, single-center study that to find out (1)The effectiveness and safety of toripalimab combined with platinum-doublet chemotherapy as a preoperative neoadjuvant therapy for locally advanced (stage IIB, IIIA, and resectable stage IIIB) NSCLC, (2)The best treatment time for this combination of neoadjuvant therapy before surgery, (3)The effectiveness and safety of combination of neoadjuvant therapy as salvage neoadjuvant therapy after failure of neoadjuvant chemo-only for locally advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Sign the informed consent form before starting any trial related procedure.
* 18-80 years old, male or female.
* Non-small cell lung cancer confirmed by cytology or histology. Evaluation by the researchers to confirm resectable stage IIB, IIIA or resectable stage IIIB (CT3-4N2M0) NSCLC patients without any treatment before.
* If the pathological type is adenocarcinoma, genetic testing is required.
* Newly treated patients or patients with failure of traditional preoperative neoadjuvant chemotherapy can be enrolled;
* ECOG PS 0-1.
* Good cardiac function, left ventricular ejection fraction >50%;
* Good respiratory function, able to tolerate radical resection of lung cancer;
* Bone marrow hematopoietic function is good, leukocyte> 4×10^9/l; Hemoglobin> 10g/dl; Platelet > 100×10^9/l;
* Good renal function, glomerular filtration rate>60 ml/min.
* Good liver function, Total bilirubin(TBIL)<1.5ULN, AST<2.5 ULN, ALT<3ULN;
* There must be at least one evaluable focus judged according to recist1.1 standard.

Exclusion Criteria:

small cell lung cancer confirmed by cytology or histology. Pathologic type was adenocarcinoma with EGFR gene mutation or ALK gene rearrangement.

Advanced lung cancer, or unresectable lung cancer A patient who had received preoperative neoadjuvant radiotherapy for NSCLC. Patients who have a history of active autoimmune disease or potentially recurrent autoimmune disease.

Patients with active hepatitis Allergic to study drug (Toripalimab ,cisplatin, carboplatin, paclitaxel, gemcitabine and pemetrexed) components excipients.

Patients were given antibiotics within 2 weeks. The investigator considered that the subject's comordities or other conditions may affect the compliance with the protocol or are not suitable for participating in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2023-05-21 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Major pathological response (MPR) rate | At time of surgery
  MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the pathological examination of resected specimens.

SECONDARY OUTCOMES:
Complete pathological response (pCR) rate | At time of surgery
  pCR rate is defined as the percentage of participants having no tumor cells in the pathological examination of resected specimens.
R0 surgical resection rate | At time of surgery
  No residual ratio under the microscope after surgical resection
Objective response rate (ORR) | Baseline (Prior to surgery)
  ORR is defined as the percentage of participants having a complete response or a partial response, measured by RECIST 1.1.
Adverse Events (AEs) | Approximately 2 years after the last patient registered.
  Incidence of all grade AE which has been confirmed to be correlated with neoadjuvant treatment.
Event-free survival(EFS) | Approximately 2 years after the last patient registered.
  Event-free survival was defined as the time from the first treatment to any progression of disease precluding surgery, progression or recurrence of disease after surgery, progression of disease in the absence of surgery, or death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu B, Tao Y, Zhuo M, Xu LD, Cheng X, Tao W, Xie Z, Lv C, Wang Y, Li S, Zhang S, Huang M, Wang Y, Li X, Zhu Y, Cui X, Zhou X, Han B, Zhang E, Huang YS, Chen W, Wang J, Yan S, Wu N. The role of dynamic monitoring of plasma cell-free DNA methylation in predicting pathological response in resectable stage IIB-IIIB non-small cell lung cancer: biomarker analyses from a prospective phase II trial. BMC Med. 2025 Nov 5;23(1):611. doi: 10.1186/s12916-025-04419-x. PMID 41194150
- [Derived] Tao Y, Li X, Liu B, Wang J, Lv C, Li S, Wang Y, Chen J, Yan S, Wu N. Association of early immune-related adverse events with treatment efficacy of neoadjuvant Toripalimab in resectable advanced non-small cell lung cancer. Front Oncol. 2023 May 15;13:1135140. doi: 10.3389/fonc.2023.1135140. eCollection 2023. PMID 37256186